CLINICAL TRIAL: NCT01222169
Title: Impact of Intravenous Lidocaine on Laryngeal Reflex Responses in Pediatric Patients Anesthetized With Propofol
Brief Title: Laryngeal Reflex Study Under Propofol Anesthesia: Effect of Intravenous Lidocaine
Acronym: LR6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Erb (Other)
Responsible Party: Sponsor-Investigator, Thomas Erb, Prof. Dr. Thomas O. Erb, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UKBB_ANA_LR 6
Record Dates: First submitted 2010-09-23; First posted 2010-10-18 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Laryngospasm
Keywords: Anesthesia; Children; Larynx
MeSH Terms: conditions — Laryngismus; Laryngeal Diseases | interventions — Propofol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- larynx assessment under stimulation (Experimental)
  Interventions: Drug: NaCl 0,9%
- Larynx assessment under stimulation (Placebo Comparator)
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: NaCl 0,9% — Propofol 3micrgr/ml (TCI plasma concentration) and NaCl 0,9% 2min. and 10min. application
  Other Names: Propofol; Disoprivan; Recofol; Natriumchlorid

SUMMARY:
To describe respiratory and laryngeal responses to laryngeal stimulation during propofol anesthesia in children. To determine whether the co-administration of lidocaine blunts these reflex responses. The outcome of primary interest is the reflex laryngospasm.

Hypotheses:

I: The severity of laryngospasm evoked by laryngeal stimulation is reduced 2 min. after iv. administration on 2mg/kg lidocaine in pediatric patients anesthetized with propofol (3mcg/ml).

II:The incidence of laryngospasm elicited by controlled stimulation 10min. after iv. administration of lidocaine is equivalent to the response before the administration of lidocaine.

DETAILED DESCRIPTION:
Based on our previous work assessing the laryngeal reflex responses in children, the use of propofol appears to be promising regarding a low incidence of laryngospasm. Compared with a sevoflurane-based anesthesia, the incidence was found to be significantly lower, but there is a high incidence of other reflex responses, such as coughing and expiration reflexes. The use of lidocaine has been advocated to reduce the incidence of laryngospasm in anesthetized children. However, based on clinical studies its effectiveness in the prevention or attenuation of laryngospasm is controversial.

In a previous work using a established stimulation model (stimulating the laryngeal mucosa with a small amount of distilled water under direct fiberbronchoscopic observation), we observed a risk reduction of 60% of laryngospasm 2min. after the application of 2mg/kg bolus of lidocaine. This effect had already diminished after 10 min.

The laryngeal reflex responses differ largely in children anesthetized with either inhalational anesthetics or with propofol. The impact iv administered lidocaine on laryngeal and respiratory reflex responses in children anesthetized with propofol has not been assessed, although this combination might result in a profound suppression of laryngeal reflex responses.

ELIGIBILITY:
Inclusion Criteria:

* 25 - 84 months
* gender: female / male
* elective surgery or diagnostic procedure requiring general anesthesia

Exclusion Criteria:

* respiratory infection within the last 2 weeks
* reactive airway disease under therapy
* cardiovascular disease
* neuromuscular disease
* positive family history of malignant hyperthermia
* known hypersensitivity to the investigational medical product
* Participation in another study
* Inability of the parents to read and understand the participant's information

Ages: 25 Months to 84 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Occurence of laryngospasm (defined as complete adduction of vocal cords and/or fals cords) with apnea lasting >10sec after laryngeal stimulation | 10 min.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas O Erb, Professor MD, Principal Investigator — University children's hospital beider Basel
Locations (1):
- University children's hospital beider Basel, Basel, Switzerland